CLINICAL TRIAL: NCT02450292
Title: Retrospective CT Imaging of BioComposite Interference Screw in Patients Undergoing Anterior Cruciate Ligament Reconstruction With Bone-Patellar Tendon-Bone Graft
Brief Title: Retrospective CT Imaging of BioComposite Interference Screw With BTB
Status: Completed | Type: Observational
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Marc Fineberg, Chief of Sports Medicine, Associate Professor of Clinical Orthopaedics, State University of New York at Buffalo
Other Study IDs: 758594-1
Record Dates: First submitted 2015-05-18; First posted 2015-05-21 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: ACL Tear
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Bioabsorbable screw fixation

SUMMARY:
The purpose of this study is to examine the long-term appearance and resorption rate of biocomposite screws used during ACL reconstruction on X-ray and computed tomography (CT).

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-50
* Patients who underwent primary ACL reconstruction performed by one of the study investigators at least 5 years ago
* Isolated ACL tear
* Type of graft used was bone-patellar tendon-bone autograft
* Type of screw used to attach graft to the tibia and/or femur was a BioComposite interference screws (Arthrex, Inc.)
* No degenerative joint disease on preoperative X-rays (> 50% joint space loss, presence of osteophytes)

Exclusion Criteria:

* Revision ACL reconstructions
* Types of grafts other than bone-patellar tendon-bone autograft were used
* ACL tear with concomitant pathology
* Degenerative joint disease on preoperative X-ray (> 50% joint space loss, presence of osteophytes)
* Metal or other types of bioabsorbable screws other than BioComposite interference screws (Arthrex, Inc.) were used
* ACL reconstruction performed less than 5 years ago
* Pregnancy
* Greater than Grade 2 laxity of other ligaments
* No additional fixation

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults aged 18+ who had an anterior cruciate ligament (ACL) reconstruction about 5 years ago performed by one of the study investigators.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2015-09; Primary Completion 2016-02 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Screw resorption | 5 years
  Evaluated on X-ray and CT

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fineberg, MD, Principal Investigator — University at Buffalo